CLINICAL TRIAL: NCT03596580
Title: Clinical Validation of a Screening Tool to Assess Dehydration in Older Population
Brief Title: Validation of a Screening Tool to Assess Dehydration in Hospitalized Older Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: GDST-M
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Dehydration Hypertonic; Aged
Keywords: Screening tool

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood urea, glucose, sodium and potassium; skin and mouth hydration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dehydrated participants: 125 participants ≥ 65 years of age at the moment of the interviews; hospitalized in General Medicine; osmolarity ≥ 296 mOsm/L
- Hydrated participants: 97 participants ≥ 65 years of age at the moment of the interviews; hospitalized in General Medicine; osmolarity < 296 mOsm/L

SUMMARY:
The study aims to verify the sensitivity and specificity of a tool to assess the state of hydration of the older person to identify those at risk of dehydration.

DETAILED DESCRIPTION:
Dehydration is the result of insufficient ﬂuid intake and can be consequent to an alteration of thirst mechanisms or ﬂuid loss from the intestinal and respiratory tracts. The use of diuretics can lead to dehydration too. The risk of dehydration induced by acute or chronical diseases is increased in older people because of the reduced capacity to maintain a proper fluid balance. Lower muscle mass, reduced kidney function, physical and cognitive disabilities, blunted thirst, and polytherapy are recognized as main factors for dehydration risk in older people.For these reasons, coordinated efforts are necessary to develop comprehensive assessment tool to monitor hydration in hospitalised older adults. We need to develop a pathway of screening to detect early stage dehydration in older patients in order to correct it precociously. Presently, no standardized clinical dehydration assessment method exists and there are relatively few papers investigating hydration status. A new tool was created: the Geriatric Dehydration Screening Tool - Modified doesn't require laboratory parameters, and thus its use is feasible outside hospital settings. The aim of this study is to evaluate the diagnostic accuracy of the Geriatric Dehydration Screening Tool - Modified in the assessment of the hydration status of hospitalized older population.

ELIGIBILITY:
Inclusion Criteria:

* Complete blood tests: Urea, Glucose, Sodium, Potassium reported not more than 24 hours before the observation;
* Absence of known cognitive impairments (Mini-Mental State Examination > 24).

Exclusion Criteria:

* Age < 65;
* Mini-Mental State Examination < 24.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study will concern people aged 65 or over, admitted to the medical departments of the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico. Critical, pediatric and psychiatric areas are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | baseline
  The diagnostic accuracy of Geriatric Dehydration Screening Tool-Modified in detecting dehydrated older people, compared to the standard reference (serum osmolarity)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vivanti A, Harvey K, Ash S. Developing a quick and practical screen to improve the identification of poor hydration in geriatric and rehabilitative care. Arch Gerontol Geriatr. 2010 Mar-Apr;50(2):156-64. doi: 10.1016/j.archger.2009.03.003. Epub 2009 Apr 23. PMID 19395070
- [Background] Rodrigues S, Silva J, Severo M, Inacio C, Padrao P, Lopes C, Carvalho J, do Carmo I, Moreira P. Validation analysis of a geriatric dehydration screening tool in community-dwelling and institutionalized elderly people. Int J Environ Res Public Health. 2015 Mar 2;12(3):2700-17. doi: 10.3390/ijerph120302700. PMID 25739005
- [Background] Hooper L, Abdelhamid A, Attreed NJ, Campbell WW, Channell AM, Chassagne P, Culp KR, Fletcher SJ, Fortes MB, Fuller N, Gaspar PM, Gilbert DJ, Heathcote AC, Kafri MW, Kajii F, Lindner G, Mack GW, Mentes JC, Merlani P, Needham RA, Olde Rikkert MG, Perren A, Powers J, Ranson SC, Ritz P, Rowat AM, Sjostrand F, Smith AC, Stookey JJ, Stotts NA, Thomas DR, Vivanti A, Wakefield BJ, Waldreus N, Walsh NP, Ward S, Potter JF, Hunter P. Clinical symptoms, signs and tests for identification of impending and current water-loss dehydration in older people. Cochrane Database Syst Rev. 2015 Apr 30;2015(4):CD009647. doi: 10.1002/14651858.CD009647.pub2. PMID 25924806